CLINICAL TRIAL: NCT00239798
Title: A 24-month Extension of a One-year, Multicenter, Double Blinded Double Dummy, Randomized Study to Evaluate the Safety and Efficacy of Two Doses of FTY720 Combined With Full-dose Cyclosporine, USP [Modified] (Novartis Brand) and Steroids Versus Mycophenolate Mofetil Combined With Full-dose Cyclosporine, USP [Modified] (Novartis Brand) and Steroids, in Adult de Novo Renal Transplant Recipients
Brief Title: Efficacy and Safety of FTY720 in de Novo Adult Renal Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFTY720A2218E1
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Renal Transplantation
Keywords: Transplantation, kidney, organ transplant
MeSH Terms: interventions — Fingolimod Hydrochloride

INTERVENTIONS:
Drug: FTY720

SUMMARY:
This study will evaluate the safety and efficacy of FTY720 combined with cyclosporine and corticosteroids in patients receiving a kidney transplant.

ELIGIBILITY:
Inclusion Criteria

* Patients who have completed the 12 Month visit of the Core trial either on or off study drug.
* Female capable of becoming pregnant are required to have a medically approved method of birth control until 3 Month after study medication was stopped.

Exclusion Criteria

- None

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 255
Dates: Start 2004-11; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
IA, IB, IIA, IIB, III, or humoral acute rejection diagnosed by biopsy according to Banff 97 criteria within 36 months post transplant
Permanent resumption of dialysis within 36 months post transplant
Surgical removal of graft within 36 months post transplant
Death within 36 months post transplant
Withdrawal of consent, death, or lost to follow up within 36 months post transplant
Serum creatinine, and estimated creatinine clearance within 36 months post transplant
FEV1 , FVC, FEV1/FVC, DLCO and FEF 25%-75% within 36 months post transplant
Absolute lymphocyte count within 36 months post transplant

SECONDARY OUTCOMES:
IA, IB, IIA, IIB, III, or humoral rejection diagnosed by biopsy according to Banff 97 criteria at Month 24 and Month 36 post-transplant
Permanent resumption of dialysis at Month 24 and Month 36 post-transplant
Surgical removal of graft at Month 24 and Month 36 post-transplant
Death at Month 24 and Month 36 post-transplant
Withdrawal of consent, death, or lost to follow up at Month 24 and Month 36 post-transplant
Serum creatinine, and estimated creatinine clearance at Month 24 and Month 36 post-transplant
FEV1 , FVC, FEV1/FVC, DLCO and FEF 25%-75% at Month 24 and Month 36 post-transplant
Absolute lymphocyte count at Month 18, 24, 30 and 36

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis

REFERENCES:
- [Result] Tedesco-Silva H, Szakaly P, Shoker A, Sommerer C, Yoshimura N, Schena FP, Cremer M, Hmissi A, Mayer H, Lang P; FTY720 2218 Clinical Study Group. FTY720 versus mycophenolate mofetil in de novo renal transplantation: six-month results of a double-blind study. Transplantation. 2007 Oct 15;84(7):885-92. doi: 10.1097/01.tp.0000281385.26500.3b. PMID 17984842